CLINICAL TRIAL: NCT07315503
Title: An Open-label Study to Evaluate the Safety and Efficacy of GC012F in Patients With Difficult-to-Treat (D2T) Rheumatoid Arthritis.
Brief Title: An Open-label Study of GC012F in Rheumatoid Arthritis.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025116
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis;CAR-T cell therapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: The study plans to enroll a total of 9 evaluable subjects; GC012F will be administered at the starting dose of 2 × 10^5 CAR-T cells/kg. The first 6 subjects will be randomized in a 1:1 ratio after apheresis to the LD cohort (receiving GC012F infusion following lymphodepletion) or the LD-free cohort (directly receiving GC012F infusion without lymphodepletion). After the DLT observation period, i.e., a minimum of 28 days of following GC012F infusion, is completed for all 6 subjects, all available data (including PK, PD, safety, efficacy, and biomarker data) obtained from the treatment period will be reviewed to determine the conditioning regimen and dose for subsequent evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LD and GC012F CAR-T Cell Injection (Experimental): The first 6 subjects will be randomized in a 1:1 ratio after apheresis to the LD cohort or the LD-free cohort，in the LD cohort subject will receiving GC012F infusion following lymphodepletion,For the subsequent 3 patients, whether to perform pretreatment and the dosage of the study drug will be determined after evaluating the first 6 patients.
- GC012F CAR-T Cell Injection (Experimental): The first 6 subjects will be randomized in a 1:1 ratio after apheresis to the LD cohort or the LD-free cohort，in the LD-free cohort the subject will directly receiving GC012F infusion without lymphodepletion,For the subsequent 3 patients, whether to perform pretreatment and the dosage of the study drug will be determined after evaluating the first 6 patients.
  Interventions: Drug: GC012F CAR-T Cell Injection

INTERVENTIONS:
Drug: LD and GC012F CAR-T Cell Injection — Subjects will receive cyclophosphamide 200 to 300 mg/m2 and fludarabine 20 to 30 mg/m2 once daily for 3 days either on Days -5, -4 and -3 or on Days -4, -3 and -2 prior to CAR-T cell infusion.
  Other Names: cyclophosphamide; fludarabine
Drug: GC012F CAR-T Cell Injection — the LD-free cohort ，directly receiving GC012F infusion without lymphodepletion.
  Arms: GC012F CAR-T Cell Injection

SUMMARY:
This is An Open-label Study to Evaluate the Safety and Efficacy of GC012F in Patients with Difficult-to-Treat (D2T) Rheumatoid Arthritis.

DETAILED DESCRIPTION:
This is an open-label, early exploratory clinical study designed to evaluate the safety and efficacy as well as PK and PD profiles of GC012F infusion with or without lymphodepletion in patients with D2T RA.

The study consists of a screening period, apheresis day(s), a baseline period, a period of lymphodepletion conditioning (applicable to subjects in the lymphodepletion cohort [LD cohort] and to those in the lymphodepletion-free cohort [LD-free cohort] who decide to undergo lymphodepletion and receive a second dose of GC012F infusion), a period of CAR-T cell infusion, and a follow-up period.

Eligible subjects will undergo apheresis and receive infusion after CAR-T product manufacturing is completed. Subjects in the LD cohort will receive lymphodepletion conditioning with fludarabine and cyclophosphamide prior to CAR-T cell infusion. All subjects will be assessed prior to cell infusion, and those meeting infusion criteria will receive CAR-T cell infusion.

The study plans to enroll a total of 9 evaluable subjects; GC012F will be administered at the starting dose of 2 × 105 CAR-T cells/kg. The first 6 subjects will be randomized in a 1:1 ratio after apheresis to the LD cohort (receiving GC012F infusion following lymphodepletion) or the LD-free cohort (directly receiving GC012F infusion without lymphodepletion). After the DLT observation period, i.e., a minimum of 28 days of following GC012F infusion, is completed for all 6 subjects, all available data (including PK, PD, safety, efficacy, and biomarker data) obtained from the treatment period will be reviewed to determine the conditioning regimen and dose for subsequent evaluation. Then, the selected conditioning regimen and dose will be continuously investigated in the subsequent study, with doses being selected based on existing data and adjusted according to emerging data. If GC012F expansion is not detected after infusion in subjects of LD-free cohort, lymphodepletion and a second dose of GC012F infusion may be considered; the proposed dose for the second infusion is 2 × 105 CAR-T cells/kg. The second dose of infusion will not be included in DLT evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 1) Capable of signing the informed consent form and willing and able to comply with study procedures;
* 2) Age ≥ 18 years (or the local legal age of consent in the region where the study is conducted) and ≤ 75 years at the time of signing the informed consent form;
* 3) Women of childbearing potential (WOCBP) (women who have undergone hysterectomy or have been postmenopausal for at least 2 years are not considered to be of childbearing potential) must:
* a) Have a negative serum or urine beta-human chorionic gonadotropin (β-hCG) pregnancy test result as confirmed by the investigator during screening, as the study drug may pose potential risks or unknown effects to the fetus;
* b) Agree to avoid breastfeeding during the study and for at least 2 years after GC012F infusion, or until CAR-T cells become undetectable by two consecutive assessments using flow cytometry (whichever occurs later);
* 4) Male subjects with female partners of childbearing potential and female subjects of childbearing potential must agree to use effective contraceptive methods (such as oral contraceptives, intrauterine devices, or condoms) from the start of screening and for at least 2 years following GC012F infusion, or until CAR-T cells become undetectable by two consecutive assessments using flow cytometry (whichever occurs later); Male subjects must agree to use condoms during sexual activity with pregnant women or women of childbearing potential for at least 2 years following GC012F infusion, even if they have undergone successful vasectomy;
* 5) Able to establish venous access required for apheresis, with no contraindications to apheresis.
* 6) Laboratory test results during screening must meet the following criteria (excluding criteria specific to the disease under study):

Organ and bone marrow function:

* Absolute neutrophil count ≥ 1.0 × 109/L (no growth factor support within 7 days prior to laboratory tests);
* Absolute lymphocyte count ≥ 0.5 × 109/L;
* Hemoglobin ≥ 80 g/L (no pre-transfusion of red blood cells within 7 days prior to laboratory tests);
* Platelet count ≥ 50 × 109/L (no pre-transfusion within 7 days prior to laboratory tests);
* Serum immunoglobulin G (IgG) ≥ 500 mg/dL;
* Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, prothrombin time (PT) ≤ 1.5 × ULN;
* Adequate renal, hepatic, pulmonary, and cardiac function, defined as:
* i. Serum alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 3 × ULN;
* ii. Total bilirubin (TBIL) < 2 × ULN (for subjects with Gilbert's syndrome, direct bilirubin [DBIL] ≤ 1.5 × ULN);
* iii. Creatinine ≤ 2 mg/dL or creatinine clearance (estimated using the Cockcroft-Gault formula) ≥ 60 mL/min;
* iv. Left ventricular ejection fraction (LVEF) ≥ 45% obtained with echocardiography (ECHO) or multigated acquisition (MUGA) scans (performed within ≤ 8 weeks prior to apheresis), no clinically significant evidence of pericardial effusion by ECHO (except for cases caused by RA), and no clinically significant abnormal electrocardiogram findings;
* v. Baseline oxygen saturation > 92% in room air;
* 7) Meet the 2010 ACR-EULAR classification criteria for RA;
* 8) Meet the EULAR 2021 definition of D2T-RA
* i. Those who have been treated according to EULAR guidelines and failed to respond to csDMARDs after failure of at least 2 bDMARDs/tsDMARDs with different mechanisms of action (unless contraindicated);
* ii. Signs suggestive of active/progressive disease, defined as ≥1 of:
* a. Moderate or higher disease activity (determined using a validated composite scale including joint counts, such as DAS28-ESR > 3.2 or CDAI > 10);
* b. Clinical manifestations (including acute phase reactants and radiographic findings) and/or symptoms (joint-related or others) indicating disease activity;
* c. Inability to taper or discontinue glucocorticoids (<7.5 mg/day prednisone or equivalent);
* d. Rapid radiographic progression (with or without signs of active disease);
* e. Disease control appears adequate by the above criteria but RA symptoms still result in reduced quality of life;
* iii. Rheumatologist and/or patient considers management of symptoms and/or manifestations to be problematic;
* 9) Failure of at least 1 csDMARD and at least 2 tsDMARDs/bDMARDs (defined as insufficient response after at least 3 months of treatment);
* 10) Presence of ≥ 6 swollen joints (based on 66-joint count) and ≥ 6 tender joints (based on 68-joint count);
* 11) A DAS28-ESR or DAS28-CRP > 3.2;
* 12) Positive for both RF and ACPA.

Exclusion Criteria:

* 1) Receipt of any other investigational drug within 4 weeks prior to signing the ICF, or the ICF signing date falls within 5 half-lives after the last dose of the investigational drug during subjects' recent participation in a clinical study (whichever is longer);
* 2) Uncontrolled and/or infection requiring hospitalization or intravenous antimicrobial therapy (fungal, bacterial, viral, or other infections) within 4 weeks prior to screening. Subjects with simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis who respond to the current therapy may be enrolled;
* 3) Active tuberculosis or inadequately treated latent tuberculosis prior to or during screening;
* 4) History of severe hypersensitivity or allergy;
* 5) History of severe immediate allergic reaction to any drug used in this study, including GC012F and its excipients (including dimethyl sulfoxide), fludarabine and cyclophosphamide (applicable only to subjects who plan to receive lymphodepletion), tocilizumab, or any component of the study drug, or presence of any contraindication, life-threatening allergy, hypersensitivity, or intolerance to these agents;
* 6) Those who have inflammatory bowel disease requiring treatment or any clinically significant gastrointestinal disease within the past 5 years;
* 7) Primary immunodeficiency;
* 8) Cardiac insufficiency or clinically significant cardiac disease, including:
* a) New York Heart Association (NYHA) functional class III or IV congestive heart failure within 6 months prior to enrollment;
* b) Acute coronary syndrome/myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), or coronary artery bypass grafting (CABG) within ≤ 6 months prior to enrollment, or any other clinically significant cardiac disease (including uncontrolled congestive heart failure), or planned revascularization intervention (subjects with stable cardiac disease who meet the inclusion criteria may be enrolled);
* c) Clinically significant arrhythmias (such as ventricular tachycardia, patients with atrial fibrillation/flutter with well-controlled ventricular rate [average heart rate at rest< 100 bpm] may be eligible at the investigator's discretion), QTc interval corrected by Fredericia formula > 450 ms in males or > 470 ms in females, complete left bundle branch block, high-degree atrioventricular (AV) block, or unexplained syncope at screening not attributable to vasovagal response or dehydration;
* d) Non-ischemic dilated cardiomyopathy, hypertrophic cardiomyopathy, cardiac amyloidosis, or sarcoidosis, clinically significant aortic valve stenosis, or severe aortic/mitral valve incompetence;
* e) History of severe non-ischemic cardiomyopathy;
* f) Uncontrolled hypertension.
* 9) History of severe respiratory disease or active severe respiratory disease, including moderate or more severe asthma or chronic obstructive pulmonary disease (COPD), interstitial lung disease, or pulmonary fibrosis;
* 10) Presence of or history of liver cirrhosis;
* 11) Presence of any active malignancy or history of malignancy within 5 years prior to screening, with the exception of: early-stage tumors that have received curative treatment (carcinoma in situ or stage 1 tumor with depth < 1 mm and no lymph node involvement, non-ulcerated primary melanoma), basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in situ, or ductal carcinoma in situ of the breast that has received potentially curative treatment;
* 12)Presence of clinically significant bleeding symptoms or definite bleeding tendency within 6 months prior to screening, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophilia, coagulopathy, splenomegaly), or are receiving anticoagulant therapy or concomitant antiplatelet agents; Note: Subjects with abnormal coagulation that meets any of the following criteria must be excluded: international normalized ratio (INR) > 1.5, prothrombin time (PT) > 14 seconds, partial thromboplastin time (PTT) > 45 seconds;
* 13) Clinically significant arterial or venous thrombotic events such as cerebrovascular disorders (cerebral hemorrhage, cerebral infarction, etc.), deep venous thrombosis, and/or pulmonary embolism within 6 months prior to screening;
* 14) Hematologic disorders: history of cytopenia consistent with myelodysplastic syndrome (MDS) diagnosis; history of sickle cell anemia or other hemoglobinopathies;
* 15) Severe underlying diseases, such as:
* a) Dementia or altered mental status with clinically evidence;
* b) History of any other central nervous system disease or neurodegenerative disorder, such as epilepsy, seizure, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, or psychiatric disorders;
* c) Psychiatric disorders or psychosocial conditions that may pose unacceptable risk to patients;
* 16) Any of the following positive test results:
* a) Positive for human immunodeficiency virus (HIV) antibodies;
* b) Hepatitis B surface antigen (HBsAg) positive; or hepatitis B core antibody (HBcAb) positive with hepatitis B virus (HBV) DNA above the detection limit;
* c) Hepatitis C virus (HCV) antibody-positive with HCV RNA above the detection limit;
* d) Treponema pallidum antibody-positive; The immunosuppression included in this study may pose unacceptable risks; subjects with active HIV, hepatitis B (HBsAg-positive), or hepatitis C virus (HCV antibody-positive) are excluded. Subjects with a history of hepatitis B or hepatitis C infection are allowed, provided that quantitative PCR and/or nucleic acid testing show viral loads below the detection limit. Hepatitis B surface antibodies following hepatitis B vaccination is not considered as evidence of prior infection.
* 17) Splenectomy within 12 months prior to signing the ICF;
* 18) Prior receipt of CD19 and/or BCMA-targeted therapy or any antigen-targeted CAR-T cell therapy;
* 19) Major surgery within 8 weeks prior to signing the ICF or planned surgery during the study (except for subjects scheduled for local anesthesia surgery, provided that the surgery will not be performed within 2 weeks after infusion);
* 20) History of solid organ transplantation;
* 21) Prior bone marrow/autologous hematopoietic stem cell transplantation or total lymphoid irradiation;
* 22) Pregnant women or lactating women who do not agree to discontinue breastfeeding, male or female subjects who plan to have children during the study or within 2 years after receiving study treatment;
* 23) Any condition prior to screening that, in the investigator's judgment, may compromise subject safety, interfere with interpretation of study results, or impede subject participation or protocol compliance.
* 24) History or current diagnosis of inflammatory joint diseases other than RA (including but not limited to: gout, systemic lupus erythematosus, psoriatic arthritis, axial spondyloarthritis [including ankylosing spondylitis and non-radiographic axial spondyloarthritis], reactive arthritis, overlap connective tissue diseases, scleroderma, polymyositis, dermatomyositis, fibromyalgia [with current active symptoms], or any arthritis with onset before age 17). History of secondary Sjögren's syndrome is permitted.
* 25) Diagnosis of Felty's syndrome;
* 26) Prednisone > 10 mg/day or equivalent dose within 1 week prior to apheresis;
* 27) Leflunomide use within 4 weeks prior to apheresis (Note: it is recommended that a leflunomide washout procedure should be initiated following the corresponding labeling);
* 28) Use of other conventional synthetic disease-modifying antirheumatic drugs (csDMARDs) within 1 week prior to apheresis;
* 29) Use of targeted synthetic disease-modifying antirheumatic drugs (tsDMARDs) within 2 weeks prior to apheresis;
* 30) Receipt of CD20-targeted therapy within 6 months prior to apheresis;
* 31) Use of other biological disease-modifying antirheumatic drugs (bDMARDs) within 6 weeks prior to apheresis;
* 32) Use of opioid medications within 1 week prior to apheresis;
* 33) Receipt of live attenuated vaccine within 4 weeks prior to apheresis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2041-01-15 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) Rate | 28 days
  DLT is defined as an AE that occurs within 28 days of GC012F CAR-T product reinfusion.DLT will be evaluated according to NCI-CTCAE V5.0 criteria.
Adverse Events （AEs）、Serious (SAE)、Adverse Event of Special Interest(AESI) Rate | Up to 15 years from treatment discontinuation
  Proportion of subjects experiencing AE within 15 years after infusion of GC012F CAR-T cell injection.

SECONDARY OUTCOMES:
GC012F T cell count in peripheral blood (Pharmacokinetic evaluation indicators) | Up to 15 years from treatment discontinuation
  maximum observed blood concentration, time to maximum observed blood concentration, area under the blood concentration-time curve from time 1 to 29 days after infusion, last observed measurable concentration, and time to last observed measurable CAR-T cell concentration.
GC012F CAR gene copy number in peripheral blood (Pharmacodynamic evaluation indicators,) | Up to 15 years from treatment discontinuation
  Observe blood the highest concentration of the CAR gene copy number
Changes in the concentration of soluble B-cell maturation antigen (BCMA) in peripheral blood | Up to 15 years from treatment discontinuation
  Observe blood the highest concentration of the BCMA
Quantification of cytokines Changes in peripheral blood | Up to 15 years from treatment discontinuation
  Observe blood the highest Quantification of the cytokines
Quantification of immunoglobulins (Ig) Changes in peripheral blood | Up to 15 years from treatment discontinuation
  Observe blood the highest Quantification of the immunoglobulins (Ig)
Changes in anti-citrullinated protein antibody (ACPA) levels | Up to 48 weeks after randomization
  Percentage of subjects who experience seroconversion from anti-citrullinated protein antibody (ACPA)-negative to ACPA-positive at Weeks 4, 12, 24, and 48;Change in the ACPA concentration over time;Change in levels of ACPA isotypes (including anti-CCP, anti-AKA, anti-APF).
Changes in rheumatoid factor (RF) concentration in peripheral blood | Up to 48 weeks after randomization
  Observe blood the highest concentration of rheumatoid factor;Percentage of subjects with rheumatoid factor (RF) seroconversion at weeks 4, 12, 24, and 48
Percentage of subjects developing antibodies against GC012F | Up to 15 years from treatment discontinuation
  Proportion of subjects experiencing against GC012F within 15 years after infusion of GC012F CAR-T cell injection.
Percentage of subjects achieving DAS28-CRP remission, DAS28-ESR remission at week 4, 12,24, and 48 | Up to 48 weeks after randomization
  Proportion of subjects in remission using definition: DAS28-CRP<2.6 Disease Activity Score-28 with C-Reactive Protein (DAS28-CRP) describes severity of rheumatoid arthritis using clinical and laboratory data, specifically CRP.
  Proportion of subjects in remission using definition: DAS28-ESR<2.6 Disease Activity Score-28 with Erythrocyte Sedimentation Rate (DAS28-ESR) describes severity of rheumatoid arthritis using clinical and laboratory data, specifically ESR.
Percentage of subjects achieving American College of Rheumatology (ACR) 20/50/70 response at Weeks 4, 12, 24, and 48 | Up to 48 weeks after randomization
  ACR response is scored as a percentage improvement, comparing disease activity at two discrete time points
Percentage of subjects achieving Boolean2.0 remission at Weeks 4, 12, 24, and 48 | Up to 48 weeks after randomization
  Boolean criteria of remission are : number of tender and swollen joint, visual analogue scale for global health and CRP all ≤1
Percentage of subjects achieving Clinical Disease Activity Index (CDAI) remission at Weeks 4, 12, 24, and 48 | Up to 48 weeks after randomization
  Clinical Disease Activity Index (CDAI) is a useful clinical composite score. It's the sum of 4 parameters : Swollen 28-Joint + Tender 28-Joint Count + Patient Global disease Activity + Evaluator's Global disease Activity.
Percentage of subjects achieving Simplified Disease Activity Index (SDAI) remission at Weeks 4, 12, 24, and 48 | Up to 48 weeks after randomization
  Score Disease Activity Index (SDAI) is the sum of 5 parameters: the number of painful joints and synovitis (28 joints are tested) the global assessment of the patient and the therapist on a visual

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, China, Tianjin, China